CLINICAL TRIAL: NCT05865925
Title: A Multicenter Phase I/II Clinical Study to Evaluate the Safety and Primary Efficacy of LY01616 (Irinotecan Hydrochloride and Floxuridine Liposome Injection) in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics (PK), and Primary Clinical Efficacy of LY01616 in Patients With Advanced Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LY01616/CT-CHN-101
Record Dates: First submitted 2023-04-25; First posted 2023-05-19 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- LY010616(30 mg/m2) (Experimental): 30 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616
- LY010616(60 mg/m2) (Experimental): 60 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616
- LY010616(90 mg/m2) (Experimental): 90 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616
- LY010616(120 mg/m2) (Experimental): 120 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616
- LY010616(150 mg/m2) (Experimental): 150 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616
- LY010616(180 mg/m2) (Experimental): 180 mg/m2 measured by Irinotecan hydrochloride, IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter)
  Interventions: Drug: LY010616

INTERVENTIONS:
Drug: LY010616 — IV infusion was 90min (±5min), with an interval of 3 weeks between the first administration and the second administration, and once every 2 weeks thereafter
  Other Names: Irinotecan Hydrochloride and Floxuridine liposome Injection

SUMMARY:
This is a multicenter, open, dose escalation, single and multiple administration phase Ⅰ/Ⅱ clinical study to evaluate the safety, tolerability, pharmacokinetics (PK), and primary clinical efficacy of LY01616 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* 1. A signed informed consent form (ICF) from the patient or their legally authorized representative. It has fully understood and voluntarily signed the written informed consent for this study, and can comply with the requirements and restrictions listed in the informed consent;
* 2. males or females, ages ≥18 to ≤70 years；
* 3. Patients with advanced solid tumors confirmed by histopathology and/or cytology, who are ineffective or unable to tolerate standard treatment, or who have no standard effective treatment plan (preferred target tumors such as colorectal cancer, gastric cancer, esophageal cancer, pancreatic cancer, small cell lung cancer, soft tissue sarcoma, cervical cancer, etc.);
* 4. At least one measurable lesion (according to RECIST 1.1 criteria);
* 5.ECOG < 2;
* 6. Organ function meets the following criteria during screening: i.Blood routine examination: neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, hemoglobin (Hb) ≥90g/L; ii.Liver function: Total bilirubin (TBIL) ≤1.5× upper limit of normal (ULN); Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5×ULN; If liver metastasis is present, AST and ALT≤5×ULN; iii.Renal function: serum creatinine ≤1.5×ULN or creatinine clearance ≥50mL/min (Cockcroft-Gault formula).

Exclusion Criteria:

* 1. Having a malignant tumor of the brain or other malignant hematological disease;
* 2. Complicated with symptomatic brain metastasis, meningeal metastasis, spinal cord tumor invasion and spinal cord compression;
* 3. Other malignancies (except cured cervical cancer of stage IB or lower, and non-invasive basal cell or squamous cell skin cancer) within 5 years prior to screening;
* 4. Uncontrollable large pleural effusion, ascites and pericardial effusion;
* 5. Persistent or active infection requiring intravenous treatment; If there is bleeding as determined by the investigator, it is not appropriate to enroll; Fever (axillary temperature ≥38℃);
* 6. History of acute coronary syndrome, coronary revascularization, New York Heart Association (NYHA) grade ≥II cardiac dysfunction, severe unstable ventricular arrhythmias within 6 months; Or an arrhythmia requiring treatment at the time of screening;
* 7. Anti-hepatitis C virus antibody (HCV-AB) positive, anti-human immunodeficiency virus antibody (anti-HIV) positive or syphilis antibody positive, active hepatitis B [hepatitis B surface antigen (HBsAg) positive test, And peripheral blood HBV DNA titer detection ≥ 1 x 103 copies /mL or 200 IU/ mL; if HBsAg positive, and peripheral blood HBV DNA titer detection < 1 x 103 copies /mL or 200 IU/ mL, If the investigator believes that the subject's chronic hepatitis B is stable and does not increase the subject's risk, the subject will be eligible for admission];
* 8. Electrolyte disturbances with clinical significance judged by the researcher still existed before study administration;
* 9. Severe gastrointestinal disorders (such as gastrointestinal bleeding, infection, chronic enteritis, obstruction, or CTCAE grade 1 or above diarrhea) at the time of screening;lts for drug.
* 10.A past or ongoing history of neuropathy or mental disorder (including epilepsy or dementia);
* 11.Patients with other major organ diseases (such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, rheumatic immune system or metabolic and endocrine system diseases) who are not suitable for inclusion;
* 12.Homozygous mutation of UGT1A1*28 allele (UGT1A1 TA 7/7 genotype)- Only for the dose escalation phase;
* 13.Previous irinotecan treatment;
* 14.Received systemic antitumor therapy (including radiotherapy, chemotherapy or other treatment) within 4 weeks prior to the first administration of study drug;
* 15.CYP3A4 strong inducers (phenytoin or carbamazepine, barbiturates, ripfampicin, or ripapentine, hypericum perforatum, etc.) have been used in the concomitant medication or within 14 days prior to treatment with the experimental drug;
* 16.CYP3A4 strong inhibitors (clarithromycin, ketoconazole or itraconazole, indenavir, lopinavir, nafazoldone, nerfinavir, ritonavir, saquinavir, terapivir, voriconazole, etc.) have been used in the concomitant medication or within 14 days before treatment with the experimental drug;
* 17.The use of UGT1A1 strong inhibitors (azanavir, gefirozil, indinavir, etc.) within 14 days prior to the treatment with the experimental drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) . | From the initiation of study treatment to the completion of safety follow-up after the end of study treatment, up to 2 years.

SECONDARY OUTCOMES:
Area under the curve (AUC) of LY01616 | up to cycle 6nd (cycle 1st is 21 days, the other cycles are 14 days)
Maximum Concentration (Cmax) of LY01616 | up to cycle 6nd (cycle 1st is 21 days, the other cycles are 14 days)
Time of maximum concentration (Tmax) of LY01616 | up to cycle 6nd (cycle 1st is 21 days, the other cycles are 14 days)
Objective response rate (ORR) | up to 2 years
Disease control rate (DCR) | up to 2 years
Progression-free survival (PFS) | up to 2 years
Overall survival (OS); | up to 2 years
Duration of remission (DoR) | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided